CLINICAL TRIAL: NCT02680483
Title: Atrial Fibrillation Registry in Jordan
Acronym: JoAFR
Status: Terminated | Type: Observational
Why Stopped: No interested parties agreed to enroll. Poor enrolling rate. In March 2018, the study was terminated.
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Principal Investigator, Ayman J Hammoudeh, MD, FACC, Co- investigator with Munir Zaqqa, MD, FACC, Jordan Collaborating Cardiology Group
Other Study IDs: JoAFR-JCCG
Record Dates: First submitted 2016-02-08; First posted 2016-02-11 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Registry; Middle East; Jordan; risk factors; in hospital management; long term management
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AF cohort: AF consecutive patients

SUMMARY:
Prospective registry of all new comers with Atrial fibrillation

DETAILED DESCRIPTION:
12 tertiary care centers will enroll all AF comers. Details of baseline clinical, EKG, echo, and lab data will be documented for all patients. Management is according to the physicians discretion. Patients will be followed up for 1 year for clinical endpoints including cardiovascular death, stroke, heart failure, systemic embolization and bleeding.. Anticoagulants and other cardiovascular medications will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* Admission with atrial fibrillation
* developing atrial fibrillation during hospitalization for mon AF reason.
* age 18 or more years.
* patients welling to participate in the registry.

Exclusion Criteria:

* age less than 18 years.
* patients not welling to participate.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All new admissions with atrial fibrillation above the age of 18 or those who develop atrial fibrillation during hospitalization for non AF reason.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Incidence of stroke and systemic embolization and cardiovascular death | 1 year
  all ischemic and hemorrhagic strokes and embolization to any arterial bed during follow up period

SECONDARY OUTCOMES:
Number of readmission for atrial fibrillation | 1 year
  readmission for atrial fibrillation related problem other than primary such as palpitations, hypotension, syncope, or near syncope.
Number of readmission for other cardiovascular events | 1 year
  Atrial Fibrillation in Jordan: risk factors, presentations, in hospital management, long term management, clinical events in hospital and at one year

CONTACTS AND LOCATIONS:
Overall Officials: Munir Zaqqa, MD FACC, Study Director — Istishari Hospital
Locations (1):
- Istishari hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No